CLINICAL TRIAL: NCT05447130
Title: Corneal Endothelial Evaluation After Phacoemulsification in Eyes With Pseudoexfoliation Syndrome
Brief Title: Corneal Endothelium After Phacoemulsification in Pseudo Exfoliation Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Hosny Ahmed Zein, Assistant Professor, Minia University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEX2019
Record Dates: First submitted 2022-07-03; First posted 2022-07-07 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Corneal Endothelial Cell Loss; Pseudoexfoliation Syndrome
Keywords: corneal endothelial cell loss, pseudoexfoliation syndrome , cataract
MeSH Terms: conditions — Corneal Endothelial Cell Loss; Exfoliation Syndrome; Cataract | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Corneal Endothelial Evaluation after Phacoemulsification in Eyes with Pseudoexfoliation Syndrome (Experimental)
  Interventions: Procedure: phacoemulsification
- Corneal Endothelial Evaluation after Phacoemulsification in Eyes without Pseudoexfoliation (Experimental)
  Interventions: Procedure: phacoemulsification

INTERVENTIONS:
Procedure: phacoemulsification — phacoemulsification with corneal endothelial evaluation by specular microscopy

SUMMARY:
To study corneal endothelial cells changes after phacoemulsification in patients with senile cataract and pseudoexfoliation syndrome (PEX) compared with control patients with senile cataract using specular microscope.

DETAILED DESCRIPTION:
In a prospective interventional case-control study, 20 eyes with cataract and PEX and 20 control eyes with cataract without PXE were subjected to phacoemulsification and posterior chamber foldable intraocular lens implantation in Minia University Hospital and Genaidy Eye Center between March 2019 and December 2020. Specular microscopy was done preoperatively, 3 and 6 months postoperatively. Endothelium cell density (ECD), coefficient variation (CV), hexagonality, pleomorphism and corneal thickness were evaluated and compares between PXE and control eyes.

ELIGIBILITY:
Inclusion Criteria:

* senile cataract age more than 55 years

Exclusion Criteria:

* PEX with glaucoma, eyes with cornea guttata or any corneal dystrophy, zonular dehiscence, very dense nuclear cataract (cataracta nigra) history of previous ocular surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
corneal endothelial cell loss | 6 months
  corneal endothelial cell loss

CONTACTS AND LOCATIONS:
Locations (1):
- Minia University Hospital, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided